CLINICAL TRIAL: NCT02358408
Title: System Accuracy Evaluation of Karajishi Contour and Karajishi TS Blood Glucose Monitoring Systems Following ISO 15197:2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: IDT-1416-BL
Record Dates: First submitted 2015-01-26; First posted 2015-02-09 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Self-Testing

INTERVENTIONS:
Device: Blood glucose monitoring systems for self-testing
  Other Names: Karajishi Contour, Karajishi Contour TS

SUMMARY:
The study consists of 2 parts:

The objective of part 1 of this study is the performance of a short evaluation of system accuracy for 25 subjects in order to familiarize the study personnel with the study BGMS to be used during the planned evaluation of system accuracy (see IDT-1416-BL (Part 2)), ensure that the Karajishi meters are fully functioning, assure and document the accuracy of the comparison method, evaluate and validate the processes and procedures of the study methodology. The objective of part 2 of this study is the evaluation of system accuracy following ISO 15197:2013 (E), clause 6.3 in which accuracy requirements and applicable test procedures for blood glucose monitoring systems intended for self-monitoring of blood glucose by patients are stipulated.

This study will be performed for Karajishi Contour and Karajishi Contour TS (manufacturer: Bayer Healthcare Diabetes Care) with 3 reagent system lots for each BGMS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, with type 1 diabetes, type 2 diabetes or no diabetes
* For provoked blood glucose excursions due to insulin dose adjustment: Male or female with type 1 diabetes or type 2 diabetes and intensified insulin therapy or insulin pump therapy.
* Minimum age of 18 years
* Signed informed consent form
* Legally competent and capable to understand character, meaning and consequences of the study

Exclusion Criteria

* Pregnancy or lactation period
* Severe acute disease (at the study physician's discretion)
* Severe chronic disease with potential risk during the test procedures (at the study physician's discretion)
* Physical or mental constitution that compromises the subject's capability to participate in the study (at the study physician's discretion)
* Incapability of giving informed consent
* < 18 years
* Legally incompetent
* Accommodated in an institution (e.g. psychiatric clinic)
* Language barriers potentially compromising an adequate compliance with study procedures
* Dependent from investigator or sponsor
* For provoked blood glucose excursions 50 - 80 mg/dl:
* Coronary heart disease
* Condition after myocardial infarction
* Cerebral incidence
* Peripheral arterial occlusive disease
* Hypoglycemia unawareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of System Accuracy according to ISO 15197 (see description) | For each subject, the experimental phase has an expected duration of up to 6 hours
  System accuracy criteria:
  1. Following ISO 15197:2013 (E), the BGMS shall meet both of the following criteria:
     * Criterion A: 95 % of the measured glucose values shall fall within either ± 15 mg/dl (0.83 mmol/l) of the average comparison measurement result at glucose concentrations < 100 mg/dl (5.55 mmol/l) or within ± 15 % at glucose concentrations ≥ 100 mg/dl (5.55 mmol/l).
     * Each lot shall pass acceptability criterion A.
     * Criterion B: 99 % of individual glucose measured values shall fall within zones A and B of the Consensus Error Grid (CEG) for type 1 diabetes.
  2. Applying ISO 15197:2003 accuracy criteria:
     * 95 % of the measured glucose values shall fall within either ± 15 mg/dl (0.83 mmol/l) of the average comparison measurement result at glucose concentrations < 75 mg/dl (4.2 mmol/l) or within ± 20 % at glucose concentrations ≥ 75 mg/dl (4.2 mmol/l).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Germany

REFERENCES:
- [Background] Pleus S, Baumstark A, Rittmeyer D, Jendrike N, Haug C, Freckmann G. Performance of two updated blood glucose monitoring systems: an evaluation following ISO 15197:2013. Curr Med Res Opin. 2016 May;32(5):847-55. doi: 10.1185/03007995.2016.1146666. Epub 2016 Feb 23. PMID 26809001